CLINICAL TRIAL: NCT02468934
Title: A Prospective Case Series Study of SPR Peripheral Nerve Stimulation (PNS) Therapy for the Treatment of Pain Following Total Knee Arthroplasty (TKA) Utilizing Preoperative Lead Placement
Brief Title: Electrical Stimulation for the Treatment of Pain Following Total Knee Arthroplasty (TKA) Using the SPRINT System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SPR Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0141-CSP-000
Record Dates: First submitted 2015-04-22; First posted 2015-06-11 (Estimated); Results first posted 2018-09-04 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Total Knee Replacement; Total Knee Arthroplasty; Pain; Postoperative Pain; Orthopedic Disorders
Keywords: electrical stimulation; neurostimulation; neuromodulation; TKA pain; pain following total knee replacement; total knee arthroplasty
MeSH Terms: conditions — Pain; Pain, Postoperative; Musculoskeletal Diseases | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peripheral Nerve Stimulation (Experimental): All study subjects will have up to 2 Smartpatch Leads placed in their leg that underwent total knee replacement, will use the SPRINT Peripheral Nerve Stimulation (PNS) System, and will receive electrical stimulation.
  Interventions: Device: SPRINT Peripheral Nerve Stimulation (PNS) System

INTERVENTIONS:
Device: SPRINT Peripheral Nerve Stimulation (PNS) System — The SPRINT System is an Investigational Device which delivers mild electrical stimulation to nerves in the leg that underwent lead placement. The SPRINT System includes a small wire (called a "Lead") that is placed through the skin in the upper leg. It also includes a device worn on the body that delivers stimulation (called the SPRINT Stimulator).
  Other Names: Smartpatch; Smartpatch System; SPRINT System

SUMMARY:
The purpose of this study is to determine if electrical stimulation (small levels of electricity) can safely and effectively reduce pain following total knee replacement (or total knee arthroplasty (TKA)). This study involves a device called the SPRINT System. The SPRINT System delivers mild electrical stimulation to nerves in the leg that received the knee replacement. The SPRINT System includes a small wire (called a "lead") that is placed through the skin in the upper leg. It also includes a device worn on the body that delivers stimulation (called the SPRINT Stimulator).

ELIGIBILITY:
Key Inclusion Criteria:

* At least 21 years old
* Scheduled to undergo a primary unilateral total knee replacement procedure

Key Exclusion Criteria:

* Body Mass Index (BMI) > 40 kg/m2
* Compromised immune system based on medical history
* History of valvular heart disease
* Implanted electronic device
* Joint or overlying skin infection of the affected limb
* History of recurrent skin infections
* Bleeding disorder
* Allergy to skin surface electrodes and/or medical-grade adhesive tapes
* Pregnant

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-10-22 (Actual); Primary Completion 2017-07-17 (Actual); Study Completion 2017-07-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of California San Diego, La Jolla, California
  - Duke University Medical Center, Durham, North Carolina
  - Joint Implant Surgeons, New Albany, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began September 2015 (with first subject enrollment in October 2015) and was concluded in February 2017. Subjects were screened for the study from a pool of candidates scheduled to undergo a primary unilateral total knee replacement procedure.
Pre-assignment Details: After obtaining informed consent, subjects were evaluated for eligibility.
Groups:
- Consented Subjects: These subjects signed an informed consent form and met all eligibility criteria.
Period: Overall Study
Arm/Group | Consented Subjects
Started | 27
Enrolled/Received Leads (Subjects consented, met eligibility criteria, and continued with SPRINT Lead placement.) | 24
Underwent Total Knee Arthroplasty (Subjects consented, met eligibility criteria, received Leads, and underwent total knee arthroplasty.) | 20
Completed | 20
Not Completed | 7
Not completed — Withdrawal by Subject | 4
Not completed — Screen Failure | 3

BASELINE CHARACTERISTICS:
Population: This group includes subjects that were consented, met eligibility criteria, and received Leads.
Groups:
- Enrolled/Received Leads: This group includes subjects that were consented, met eligibility criteria, and received Leads.
Arm/Group | Enrolled/Received Leads
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24
Affected Leg [Count of Participants; unit: Participants]
  Left Leg | 10
  Right Leg | 14
Reason for Total Knee Arthroplasty (TKA) [Count of Participants; unit: Participants] — The reason that each subject was scheduled to undergo a primary unilateral total knee arthroplasty (also known as total knee replacement).
  Participants
    Osteoarthritis | 24
    Rheumatoid Arthritis | 0
    Trauma | 0
    Post-Traumatic Arthritis | 0
    Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Average Knee Pain While Walking
Description: Subjects were asked to complete daily diaries to track their average pain intensity while walking during the past 24 hours over a 7-day period on an 11-point numerical rating scale where 0 represents "No Pain" and 10 represents "Pain as bad as you can imagine." The average score for each diary period was calculated across subjects, and the mean scores for weeks 1-4 is reported.
Time Frame: Postoperative Day 0 to 28 (first 4 weeks following Total Knee Arthroplasty (TKA))
Measure: Mean (Standard Error); unit: Scores on a scale
Groups:
- Underwent Total Knee Arthroplasty (TKA): These subjects were consented and met eligibility criteria, received leads, and underwent their scheduled Total Knee Arthroplasty (TKA) procedures.
Arm/Group | Underwent Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 20
Scores on a scale | 3.8 (0.34)

2. Primary Outcome: Number of Participants That Experienced at Least One Study-Related Adverse Event
Description: At each study visit following the baseline assessment at Visit 1, subjects were questioned if any changes in their medical status or condition has occurred since their previous visit. If the subject experienced a change that was an adverse event, an Adverse Event Form was completed by the site. The number of subjects that experienced at least one study-related adverse event is reported here.
Time Frame: Total of 21 months (from when the first subjects enrolled to when the last subject completed the study)
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled/Received Leads
Number analyzed (Participants) | 24
Participants | 15

3. Secondary Outcome: Average Knee Pain Over the Last 24 Hours
Description: Subjects were asked to complete daily diaries to track their average pain intensity in the past 24 hours over a 7-day period on an 11-point numerical rating scale where 0 represents "No Pain" and 10 represents "Pain as bad as you can imagine." The average score for each diary period was calculated across subjects, and the mean score for weeks 1-4 is reported.
Time Frame: Postoperative Day 0 to 28 (first 4 weeks following Total Knee Arthroplasty (TKA))
Measure: Mean (Standard Error); unit: Scores on a scale
Groups:
- Underwent Total Knee Arthroplasty (TKA): These subjects were consented and met eligibility criteria, received leads, and underwent their scheduled Total Knee Arthroplasty procedures.
Arm/Group | Underwent Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 20
Scores on a scale | 3.5 (0.30)

4. Secondary Outcome: Average Knee Pain at Rest
Description: Subjects were asked to complete daily diaries to track their average pain intensity at rest in the past 24 hours over a 7-day period on an 11-point numerical rating scale where 0 represents "No Pain" and 10 represents "Pain as bad as you can imagine." The average score for each diary period was calculated across subjects, and the mean score for weeks 1-4 is reported.
Time Frame: Postoperative Day 0 to 28 (first 4 weeks following Total Knee Arthroplasty (TKA))
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Underwent Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 20
Scores on a scale | 2.9 (0.29)

5. Secondary Outcome: Amount of Analgesic Usage
Description: The amount and type of analgesics used by subjects was recorded in daily diaries. Narcotic usage was converted into a morphine equivalent dosage (MED), which is measured in units of morphine milligram equivalents (MME). Diaries were collected at various visits throughout the study, and for consistency, these data were translated into post-operative days. The average MED was calculated for each subject for the first 42 days (6 weeks) following surgery, and the median of these averages was determined across subjects.
Time Frame: Visit 4 (Day of Surgery) and Visits 6-11 (weeks 1-6 post-Total Knee Arthroplasty (TKA))
Population: Data was not available for: one subject during Post-op Week 1, three subjects for Weeks 2 and 4, four subjects during Weeks 3 and 5, and for seven subjects during Post-op Week 6.
Measure: Median (Inter-Quartile Range); unit: MME (Morphine Milligram Equivalents)
Arm/Group | Underwent Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 20
MME (Morphine Milligram Equivalents) | 15.9 [7.0 to 33.8]

6. Secondary Outcome: Number of Participants That Experienced at Least One Opioid-Related Side Effect
Description: Throughout the study, subjects were asked if they experienced any side effects related to opioid pain medications. The occurrences of these side effects were recorded and were not reported as Adverse Events. The number of subjects that experienced at least one opioid-related side effect at each visit is reported.
Time Frame: Visit 1 (Baseline), Visit 2 (Lead Placement), Visits 5-13 (in-hospital days through 3-months post-Total Knee Arthroplasty (TKA))
Population: Data was not collected for: eight subjects at Visit 2, two subjects at Visit 10, and one subject at Visit 12.
Measure: Count of Participants; unit: Participants
Arm/Group | Underwent Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 20
Participants
  Visit 1 (Baseline) | 7
  Visit 2 (Lead Placement): number analyzed (Participants) | 12
  Visit 2 (Lead Placement) | 1
  Visit 5 (In-Hospital) | 13
  Visit 6 (1-week Post-TKA) | 17
  Visit 7 (2-weeks Post-TKA) | 11
  Visit 8 (3-weeks Post-TKA) | 11
  Visit 9 (4-weeks Post-TKA) | 9
  Visit 10 (5-weeks Post-TKA): number analyzed (Participants) | 18
  Visit 10 (5-weeks Post-TKA) | 7
  Visit 11 (6-weeks Post-TKA) | 4
  Visit 12 (2-months Post-TKA): number analyzed (Participants) | 19
  Visit 12 (2-months Post-TKA) | 2
  Visit 13 (3-months Post-TKA) | 1

7. Secondary Outcome: Time to Achieve 90 Degrees Flexion in Affected Knee
Description: Active range of motion (AROM; no assistance from clinical staff) and passive range of motion (PROM; assisted by clinical staff) was assessed with both stimulation on and off. The time that it took subjects to achieve the milestone of 90 degrees of knee flexion in their affected leg is reported.
Time Frame: Visit 2 (Lead Placement), Visit 7 (3-weeks Post-Total Knee Arthroplasty (TKA)), Visit 11 (6-weeks Post-TKA), Visit 13 (3-months Post-TKA)
Population: Three subjects did not meet 90 degrees of flexion with stimulation on by Visit 11 (End of Treatment) for both active range of motion (AROM) and passive range of motion (PROM). Data was not collected for four subjects for PROM with stimulation on and for three subjects for AROM with stimulation on.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Underwent Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 20
days
  PROM - Stimulation Off | 40.0 [16.0 to 44.0]
  PROM - Stimulation On: number analyzed (Participants) | 13
  PROM - Stimulation On | 16.0 [15.0 to 17.0]
  AROM - Stimulation Off | 36.5 [16.0 to 44.0]
  AROM - Stimulation On: number analyzed (Participants) | 14
  AROM - Stimulation On | 16.0 [15.0 to 17.0]

8. Secondary Outcome: Timed Up and Go (TUG) Test
Description: Subjects began this test from a seated position in a standard chair and were timed while they stood up, walked to a marked point 10 feet away (at a normal, safe pace), returned to the chair, and sat down. Timed Up and Go (TUG) test times are expected to be greater immediately after surgery as compared to baseline.
Time Frame: Visit 1 (Baseline), Visit 5 (In-Hospital), Visit 7 (2-weeks Post-Total Knee Arthroplasty (TKA)), Visit 11 (6-weeks Post-TKA), Visit 13 (3-months Post-TKA)
Population: Data was not collected for two subjects at Visit 5 and another subject was physically unable to complete the test. Data was not collected for one subject at Visit 7.
Measure: Median (Inter-Quartile Range); unit: Seconds
Arm/Group | Underwent Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 20
Seconds
  Time at Visit 1 (Baseline) | 12.3 [11.0 to 14.0]
  Time at Visit 5 (In-Hospital): number analyzed (Participants) | 17
  Time at Visit 5 (In-Hospital) | 39.0 [28.0 to 52.0]
  Time at Visit 7 (2-weeks Post-TKA): number analyzed (Participants) | 19
  Time at Visit 7 (2-weeks Post-TKA) | 13.9 [11.0 to 17.0]
  Time at Visit 11 (6-weeks Post-TKA) | 10.5 [8.0 to 13.0]
  Time at Visit 13 (3-months Post-TKA) | 8.7 [7.0 to 11.0]

9. Secondary Outcome: 6 Minute Walk Test (6MWT)
Description: The total distance that a subject could walk in 6 minutes was recorded, and the mean distance was determined across subjects. 6 Minute Walk Test distances are expected to be reduced immediately after surgery as compared to baseline.
Time Frame: Visit 1 (Baseline), Visit 7 (2-weeks Post-Total Knee Arthroplasty (TKA)), Visit 11 (6-weeks Post-TKA), Visit 13 (3-months Post-TKA)
Population: One subject at Visit 1 and two subjects at Visit 7 were physically unable to complete the test. Data was not collected for an additional subject at Visit 7.
Measure: Mean (Standard Error); unit: meters
Arm/Group | Underwent Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 20
meters
  Visit 1 (Baseline): number analyzed (Participants) | 19
  Visit 1 (Baseline) | 363.0 (15.14)
  Visit 7 (2-weeks Post-TKA): number analyzed (Participants) | 17
  Visit 7 (2-weeks Post-TKA) | 289.0 (21.55)
  Visit 11 (6-weeks Post-TKA) | 365.8 (17.87)
  Visit 13 (3-months Post-TKA) | 410.3 (16.78)

10. Secondary Outcome: Fixed Distance Walk Test
Description: The amount of time it took subjects to walk a fixed distance of 20 meters was recorded.
Time Frame: Visit 1 (Baseline) and Visit 5 (In-Hospital)
Population: One subject at Visits 1 and 5 was physically unable to complete the test. Data was not collected for two additional subjects at Visit 5, and another subject walked a fixed distance greater than 20 meters during the test so their results are not comparable.
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Underwent Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 20
seconds
  Visit 1 (Baseline): number analyzed (Participants) | 19
  Visit 1 (Baseline) | 18.1 [17.0 to 22.0]
  Visit 5 (In-Hospital): number analyzed (Participants) | 16
  Visit 5 (In-Hospital) | 48.5 [44.0 to 72.0]

11. Secondary Outcome: Percent Change From Baseline on the Western Ontario McMaster University Osteoarthritis Index (WOMAC)
Description: The Western Ontario McMaster University Osteoarthritis Index (WOMAC) questionnaire consists of 24 items that evaluate pain, stiffness, and physical functional disability. Each item is scored on an 11-point numerical rating scale from 0 to 10, where higher scores indicate greater pain, stiffness, and disability. For each subject, the scores from each of the 24 items were summed to calculate the subject's total score, with a minimum score of 0 and a maximum score of 240. Percent change from baseline was calculated for each subject at each time point (i.e., value at Visit 5 vs. Baseline rating, value at Visit 7 vs. Baseline rating, value at Visit 11 vs. Baseline rating, and value at Visit 13 vs. Baseline rating). The median percent change across subjects was determined. Negative values indicate worsening since Baseline, while positive values indicate improvement from Baseline.
  Percent improvement = 100 x ([rating at each study visit]-[rating at baseline]) / [rating at baseline].
Time Frame: as for outcome 8
Population: Data was not collected for two subjects at Visit 5.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Underwent Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 20
percent change
  Visit 5 (In-Hospital): number analyzed (Participants) | 18
  Visit 5 (In-Hospital) | -2.3 [-38.3 to 22.7]
  Visit 7 (2-weeks Post-TKA) | 39.0 [-24.1 to 58.3]
  Visit 11 (6-weeks Post-TKA) | 64.5 [37.9 to 73.3]
  Visit 13 (3-months Post-TKA) | 88.5 [68.9 to 96.8]

12. Secondary Outcome: Knee Pain Interference With Daily Activities
Description: Subjects were asked to rate the degree to which their knee pain has interfered with 7 different aspects of their daily life on a scale from 0 to 10, with higher scores indicating greater interference. Those 7 scores were averaged for each subject to provide an overall pain interference score, with a possible range of 0 to 10 with higher scores indicating greater interference. The median score was then calculated across subjects.
Time Frame: as for outcome 6
Population: Data was not collected for: 10 subjects at Visit 2, two subjects at Visit 10, and one subject at Visit 12.
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Underwent Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 20
Scores on a scale
  Visit 1 (Baseline) | 4.2 [1.7 to 6.6]
  Visit 2 (Lead Placement): number analyzed (Participants) | 10
  Visit 2 (Lead Placement) | 4.4 [2.7 to 6.6]
  Visit 5 (In-Hospital) | 3.6 [3.0 to 5.2]
  Visit 6 (1-week Post-TKA) | 3.1 [2.3 to 4.8]
  Visit 7 (2-weeks Post-TKA) | 3.1 [2.1 to 5.3]
  Visit 8 (3-weeks Post-TKA) | 2.4 [1.7 to 4.5]
  Visit 9 (4-weeks Post-TKA) | 3.6 [1.8 to 5.3]
  Visit 10 (5-weeks Post-TKA): number analyzed (Participants) | 18
  Visit 10 (5-weeks Post-TKA) | 1.8 [0.8 to 3.6]
  Visit 11 (6-weeks Post-TKA) | 1.5 [0.4 to 2.6]
  Visit 12 (2-months Post-TKA): number analyzed (Participants) | 19
  Visit 12 (2-months Post-TKA) | 0.3 [0.0 to 2.4]
  Visit 13 (3-months Post-TKA) | 0.1 [0.0 to 0.3]

13. Secondary Outcome: Number of Participants Reporting Meaningful Improvement, Minimal or No Change, or Meaningful Worsening on the Patient Global Impression of Change (PGIC) Survey
Description: The Patient Global Impression of Change (PGIC) asks subjects to rate their improvement with treatment on a 7-point scale ranging from "very much worse" to "very much improved" as compared to before their knee replacement surgery. The subjects combine all the components of their experience into one overall score. Ratings of Much- or Very Much Improved are considered Meaningful Improvements; similarly, ratings of Much- or Very Much Worse are categorized as Meaningfully Worse.
Time Frame: Visits 5-13 (in-hospital through 3-months post-Total Knee Arthroplasty (TKA))
Population: Data was not collected for two subjects at Visit 5, for three subjects at Visit 10, and for one subject at Visit 12.
Measure: Count of Participants; unit: Participants
Arm/Group | Underwent Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 20
Participants
  Visit 5 (In-Hospital): number analyzed (Participants) | 18
  Visit 5 (In-Hospital): Meaningful Improvement | 3
  Visit 5 (In-Hospital): Minimal or No Change | 8
  Visit 5 (In-Hospital): Meaningfully Worse | 7
  Visit 6 (1-week Post-TKA): Meaningful Improvement | 6
  Visit 6 (1-week Post-TKA): Minimal or No Change | 11
  Visit 6 (1-week Post-TKA): Meaningfully Worse | 3
  Visit 7 (2-weeks Post-TKA): Meaningful Improvement | 6
  Visit 7 (2-weeks Post-TKA): Minimal or No Change | 11
  Visit 7 (2-weeks Post-TKA): Meaningfully Worse | 3
  Visit 8 (3-weeks Post-TKA): Meaningful Improvement | 9
  Visit 8 (3-weeks Post-TKA): Minimal or No Change | 9
  Visit 8 (3-weeks Post-TKA): Meaningfully Worse | 2
  Visit 9 (4-weeks Post-TKA): Meaningful Improvement | 5
  Visit 9 (4-weeks Post-TKA): Minimal or No Change | 13
  Visit 9 (4-weeks Post-TKA): Meaningfully Worse | 2
  Visit 10 (5-weeks Post-TKA): number analyzed (Participants) | 17
  Visit 10 (5-weeks Post-TKA): Meaningful Improvement | 8
  Visit 10 (5-weeks Post-TKA): Minimal or No Change | 9
  Visit 10 (5-weeks Post-TKA): Meaningfully Worse | 0
  Visit 11 (6-weeks Post-TKA): Meaningful Improvement | 11
  Visit 11 (6-weeks Post-TKA): Minimal or No Change | 7
  Visit 11 (6-weeks Post-TKA): Meaningfully Worse | 2
  Visit 12 (2-months Post-TKA): number analyzed (Participants) | 19
  Visit 12 (2-months Post-TKA): Meaningful Improvement | 15
  Visit 12 (2-months Post-TKA): Minimal or No Change | 3
  Visit 12 (2-months Post-TKA): Meaningfully Worse | 1
  Visit 13 (3-months Post-TKA): Meaningful Improvement | 19
  Visit 13 (3-months Post-TKA): Minimal or No Change | 1
  Visit 13 (3-months Post-TKA): Meaningfully Worse | 0

14. Secondary Outcome: Pain Catastrophizing Scale (PCS)
Description: The Pain Catastrophizing Scale (PCS) questionnaire has 13 questions that assess rumination, magnification, and helplessness. Subjects are asked to think back on painful experiences in the past and reflect on how often they had specific thoughts or feelings. Each of the 13 questions is scored on a 5-point scale where 0 represents "not at all," and 4 represents "all the time." The scores from each question were summed for each subject to provide a total PCS score, with a possible range from 0 to 52 with higher scores indicating a greater tendency to catastrophize pain (i.e. a higher score indicates a worse outcome). The median scores were then calculated across all subjects.
Time Frame: Visit 1 (Baseline), Visit 11 (6-weeks post-Total Knee Arthroplasty (TKA)), Visit 13 (3-months post-TKA)
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Underwent Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 20
Scores on a scale
  Visit 1 (Baseline) | 5.5 [0.8 to 11.3]
  Visit 11 (6-weeks Post-TKA) | 2.0 [0.0 to 6.0]
  Visit 13 (3-months Post-TKA) | 0.0 [0.0 to 2.0]

15. Secondary Outcome: Time to Meet Recovery Milestones up to Three Months Post-Total Knee Arthroplasty (TKA)
Description: Participants were queried weekly from the date of their Total Knee Arthroplasty (TKA) until they met specific, post-surgical recovery milestones. Participants were queried up through the time at which they meet each milestone or through their completion of the study, whichever came first (up to three months post-surgery).
Time Frame: From Day of Surgery through completion of milestone or 3-months from Day of Surgery, whichever came first
Population: Data were not available for climbing stairs and discharge destination for 3 subjects and for discharge criteria and clearance to drive for one. Data were not collected for clearance to work in 2 subjects, and 10 subjects were retired. Opioid cessation data were not collected for 1 subject, and 2 subjects did not cease opioids during the study.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Underwent Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 20
days
  Pain controlled without nerve block | 1.0 [0.0 to 1.0]
  Walked with assistive device | 1.0 [0.0 to 1.0]
  Walked without assistive device | 19.5 [8.5 to 38.3]
  Walked 30 meters | 1.0 [1.0 to 2.3]
  Able to climb half flight of stairs: number analyzed (Participants) | 17
  Able to climb half flight of stairs | 7.0 [3.0 to 19.0]
  Met hospital discharge criteria: number analyzed (Participants) | 19
  Met hospital discharge criteria | 1.0 [1.0 to 3.0]
  Discharged from hospital | 1.5 [1.0 to 3.0]
  Cleared to drive: number analyzed (Participants) | 19
  Cleared to drive | 28.0 [17.0 to 39.5]
  Returned to work: number analyzed (Participants) | 8
  Returned to work | 24.0 [13.8 to 34.5]
  Cessation of all opioid medications: number analyzed (Participants) | 17
  Cessation of all opioid medications | 34.0 [10.0 to 44.0]

16. Secondary Outcome: Subject Satisfaction Survey
Description: Subjects completed a sponsor-developed survey with questions pertaining to their feelings about the SPRINT Stimulation System as a method for managing post-surgical pain.
Time Frame: Visit 11 (6-weeks post-Total Knee Arthroplasty (TKA))
Population: Two subjects did not answer the question regarding the amount of time it took to feel pain relief from stimulation.
Measure: Count of Participants; unit: Participants
Arm/Group | Underwent Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 20
Participants
  Tolerated Lead placement with some/no discomfort | 17
  Reported stimulation felt comfortable/soothing | 10
  Reported immediate pain relief (0-5 minutes): number analyzed (Participants) | 18
  Reported immediate pain relief (0-5 minutes) | 8
  Would recommend stimulation therapy to a friend | 12
  Prefer stimulation therapy to pain medication use | 14
  Wanted stimulation for longer time period | 1

ADVERSE EVENTS:
Time Frame: 21 months (from the time the first subject was enrolled to when the last subjects completed the study)
Arm/Group | Enrolled/Received Leads
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 1/24
Other Adverse Events (participants affected / at risk) | 18/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled/Received Leads (N=24)
Ileus (Gastrointestinal disorders) | 1 (2) — Not study-related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled/Received Leads (N=24)
Nausea/Upset Stomach (Gastrointestinal disorders) | 2 (2) — One event was study-related, and the other was not
Agitation (General disorders) | 3 (3) — One event was study-related, and the other two were not
Common Cold (General disorders) | 1 (1) — Not study-related
Small dehiscence at Total Knee Arthroplasty (TKA) surgical site (Skin and subcutaneous tissue disorders) | 1 (1) — Not study-related
Iliotibial Band Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) — Not study-related
Pulled Hamstring (Musculoskeletal and connective tissue disorders) | 1 (1) — Not study-related
Muscle Pain/Cramping (Musculoskeletal and connective tissue disorders) | 2 (4) — Three events were study-related, and one was not
Increased Pain (Hip and Leg) (Musculoskeletal and connective tissue disorders) | 2 (3) — Two events were not study-related, and the relationship to the study was unable to be determined for the other event
Headache (Nervous system disorders) | 1 (1) — Relationship to study unable to be determined
Pain due to Stimulation (Product Issues) | 1 (1) — Study-related
Shocks at Lead Exit Site (Product Issues) | 2 (2) — Study-related
Urinary Frequency (Renal and urinary disorders) | 1 (1) — Not study-related
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) — Not study-related
Skin irritation or bruising at Lead exit site (Skin and subcutaneous tissue disorders) | 7 (8) — Study-related
Skin irritation/dermatitis from bandages (Skin and subcutaneous tissue disorders) | 3 (3) — Study-related
Skin irritation from SPRINT Pad (Skin and subcutaneous tissue disorders) | 4 (6) — Study-related
Non-specified skin irritation (Skin and subcutaneous tissue disorders) | 3 (3) — Two events were study-related, and the other one was not
Bruising (Skin and subcutaneous tissue disorders) | 1 (1) — Not study-related
Itching (Skin and subcutaneous tissue disorders) | 1 (1) — Relationship to study unable to be determined
Affected Leg Swelling (Vascular disorders) | 1 (1) — Study-related
Knee Stiffness/Decreased Range of Motion (Musculoskeletal and connective tissue disorders) | 1 (1) — Not study-related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-13): https://cdn.clinicaltrials.gov/large-docs/34/NCT02468934/Prot_SAP_000.pdf